CLINICAL TRIAL: NCT04360057
Title: The Impact of Patient Motivational Dialogue (PMD) on Patient Self-advocacy for Hand Hygiene: A Feasibility Study
Brief Title: The Impact of Patient Motivational Dialogue (PMD) on Patient Self-advocacy for Hand Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC20160369H
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hand Disinfection
Keywords: Motivation, hand hygiene

STUDY DESIGN:
Intervention Model Description: Subjects will be included from two oncology clinics, one in radiation oncology and one in chemotherapy oncology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand Hygiene education (Other)
  Interventions: Other: PMD; Other: PMDPlus

INTERVENTIONS:
Other: PMD — A script used to train the physician to engage with the patient in the topic of hand hygiene compliance used on the initial visit.
  Other Names: Patient Motivational Dialogue
Other: PMDPlus — A script used to train the physician to engage with the patient in the topic of hand hygiene compliance on follow up visits
  Other Names: Patient Motivational Dialogue Plus

SUMMARY:
This exploratory cross sectional cohort study will evaluate the feasibility and fidelity of using an innovative strategy, the Patient Motivational Dialogue (PMD)/PMDPlus that will intentionally motivate and encourage the patient toward self-advocacy for their Health Care Professional's (HCP's) hand hygeine (HH) adherence.

DETAILED DESCRIPTION:
This study will be implemented with two volunteer innovation champion physicians, one in radiation oncology and one in the chemotherapy oncology clinic. If other physicians begin to use the PMD/ PMDPlus in their clinics, the initiation will be considered a positive indication of feasibility and fidelity.

New patients will be enrolled in the study starting September 2016 until the sample size reaches 30 patients per clinic (n=60). Each patient will be followed in each clinic visit longitudinal through March 2017 or until discharged from the clinic treatment depending on which comes first. PMD will be administered in the first clinic visit followed by the PMDPlus each visit thereafter to ensure an adequate treatment dose. The PMD is estimated to take about two minutes of the initial clinic visit and the PMDPlus is estimated to take about one minute of the follow-up clinic visit.

The following steps will be taken based on the innovation decision model:

1. The PI will instruct the physicians, or designee in the use of the PMD/PMDPlus. Script cards with the PMD/PMDPlus will be provided to each physician. The physician will be instructed in use of PMD at the initial visit and the PMDPlus every follow-up clinic visit thereafter until discharge from the clinic.
2. A HCP survey will be conducted pre-intervention asking the HCP: "Has a patient or family ever ask you to clean your hands? If yes, the HCP will be asked to describe the situation.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Able to understand instructions given by physician
* Receiving care in radiation oncology clinic and/or chemotherapy clinic at Cancer Therapy Research Center at University of Texas Health Science Center (UTHSCSA)

Exclusion Criteria:

* Unable to understand instructions given by physician

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
The Impact of Patient Motivational Dialogue (PMD) on Patient Self-advocacy for Hand Hygiene | At treatment completion, an average of 4-6 months
  At the last clinic visit, the PI or research assistant will ask the patient this nominal question: "Have you ever ask your physician or your HCP to clean their hands during your visits here?" If yes, describe the circumstances. If no, describe why not. Verbal responses will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Patti G Grota, Principal Investigator — University of Texas Health at San Antonio; Tony Eng, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No